CLINICAL TRIAL: NCT04060979
Title: Prospective, Double-Blinded, Randomized, Multi-Center Study for Evaluation of Two Doses of Nitric Oxide (NO) Given Intermittently Via Inhalation to Subjects With Bronchiolitis
Brief Title: Evaluation of Two Doses of Nitric Oxide (NO) Given Intermittently Via Inhalation to Subjects With Bronchiolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIT_CP_BRONC_03.01
Record Dates: First submitted 2019-08-11; First posted 2019-08-19 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-01

CONDITIONS: Bronchiolitis Acute
MeSH Terms: interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1- NO treatment- dose 1 (Experimental): Will comprise of approximately 30 patients and will receive inhalations of dose 1 of NO combined with O2/air for 40 minutes, every 4.5 hours during the day four times a day for up to 5 days in addition to standard supportive treatment.
  Interventions: Drug: Nitric Oxide; Other: Standard Supportive treatment
- Group 2- NO treatment- dose 2 (Experimental): Will comprise of approximately 30 patients and will receive inhalations of dose 2 of NO combined with O2/air for 40 minutes, every 4.5 hours during the day four times a day for up to 5 days in addition to standard supportive treatment.
  Interventions: Drug: Nitric Oxide; Other: Standard Supportive treatment
- Group 3- Control treatment (Other): Will comprise of approximately 30 patients and will receive O2/air using the same treatment schedule and equipment as groups 1 and 2, in addition to standard supportive treatment.
  Interventions: Other: Standard Supportive treatment

INTERVENTIONS:
Drug: Nitric Oxide — Nitric Oxide given intermittently via inhalation
  Arms: Group 1- NO treatment- dose 1; Group 2- NO treatment- dose 2
Other: Standard Supportive treatment — Standard Supportive treatment (including oxygen)

SUMMARY:
Prospective, Double-Blinded, Randomized, Multi-Center Study for Evaluation of Two Doses of Nitric Oxide (NO) Given Intermittently Via Inhalation to Subjects With Bronchiolitis

The proposed study judiciously expands these observations for use of NO treatment in pediatric patients with bronchiolitis aged less than 12 months. The intermittent dosing strategy used in this study has been selected to minimize the potential for adverse effects. The inclusion of two doses in the proposed pilot study is intended to determine a dose response effect and select a dose that is optimally safe and effective. The primary endpoint evaluation of time to fit for discharge will provide an effective objective measurement for the treatment effectiveness compared to standard supportive treatment of bronchiolitis.

Primary objective:

• Assess whether Nitric Oxide (NO) administered intermittently in 2 concentrations (via inhalation for 40 minutes 4 times per day for up to 5 consecutive days) in addition to Standard Supportive Treatment (SST) shortens the recovery time of infants with bronchiolitis, compared to SST alone.

Secondary objectives:

* Time to achieve O2 saturation of ≥ 92 % sustained for at least 2 hours
* Reduction in hospital Length of Stay (LOS)
* Time to achieve mTal score of ≤ 5

Safety objectives: Characterize the safety of 2 doses of NO intermittent inhalation treatment therapy as measured by Adverse Events (AE) - number and percentage of subjects that experience AEs - and Serious Adverse Events (SAEs).

A total of 90 subjects will be enrolled into the study and randomized in a 1:1:1 ratio to receive the study treatments.

Treatment administration: Treatment blindness will be kept by designation of blinded and un-blinded team members.The blinded staff will be performing the study assessment procedures and the un-blinded team will be administering the actual treatment.

Subjects' parents/legal guardian will be contacted for a follow up phone call at days 14+5 and 30+5 from the date of enrollment of the subject into the study.

DETAILED DESCRIPTION:
Prospective, Double-Blinded, Randomized, Multi-Center Study for Evaluation of Two Doses of Nitric Oxide (NO) Given Intermittently Via Inhalation to Subjects With Bronchiolitis

Bronchiolitis is a viral disease, widely spread amongst young children with significant mortality in some cases and no specific treatment available, besides supportive treatment of O2 and hydration; therefore, there is an identified unmet medical need to develop a treatment strategy for children with bronchiolitis.

When the immune system's NO generating ability is overwhelmed or compromised, infection and disease occur. Increasing the body's ability to produce more NO through gene therapy or synthetic NO donor drugs is of interest in medicine.

NO, by itself, is an essential part of the innate defense mechanism of the human immune system which becomes up-regulated by the inducible NO synthase (iNOS) during various inflammatory conditions and during microbial and viral infections. This suggests that NO treatment in appropriate concentrations is highly relevant for children with bronchiolitis.

The two previous pilot studies conducted by Beyond Air (formerly known as AIT) found that intermittent exposure to was safe and well tolerated in pediatric subjects with acute bronchiolitis age 0-12 months and showed a trend in reduction in the length of hospitalization. The overall frequency of adverse events was found to be similar between the control and NO treated groups and intermittent exposure at 160 ppm did not result in exposure to unsafe Nitric Dioxide (NO2) levels or had a cumulative effect on MetHb levels.

The proposed study judiciously expands these observations for use of NO treatment in pediatric patients with bronchiolitis aged less than 12 months. The intermittent dosing strategy used in this study has been selected to minimize the potential for adverse effects. The inclusion of two doses in the proposed pilot study is intended to determine a dose response effect and select a dose that is optimally safe and effective. The primary endpoint evaluation of time to fit for discharge will provide an effective objective measurement for the treatment effectiveness compared to standard supportive treatment of bronchiolitis.

NO therapy can be cost effective, technologically simple and easily adaptive for use in inhaled pulmonary infections. Ultimately, therapeutic use of NO could be the initial treatment by mimicking the body's natural first line method to fight infections. Together, these results and rationale warrant the need to accelerate research of NO as a potential solution for front line treatment for bronchiolitis.

Primary objective:

• Assess whether Nitric Oxide (NO) administered intermittently in 2 concentrations (via inhalation for 40 minutes 4 times per day for up to 5 consecutive days) in addition to Standard Supportive Treatment (SST) shortens the recovery time of infants with bronchiolitis, compared to SST alone.

Secondary objectives:

* Time to achieve O2 saturation of ≥ 92 % sustained for at least 2 hours
* Reduction in hospital Length of Stay (LOS)
* Time to achieve mTal score of ≤ 5

Safety objectives: Characterize the safety of 2 doses of NO intermittent inhalation treatment therapy as measured by Adverse Events (AE) - number and percentage of subjects that experience AEs - and Serious Adverse Events (SAEs).

A total of 90 subjects will be enrolled into the study and randomized in a 1:1:1 ratio to receive the study treatments.

Treatment administration: Treatment blindness will be kept by designation of blinded and un-blinded team members.The blinded staff will be performing the study assessment procedures and the un-blinded team will be administering the actual treatment.

Subjects' parents/legal guardian will be contacted for a follow up phone call at days 14+5 and 30+5 from the date of enrollment of the subject into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects up to 12-months of age, including subjects born ≥ 28 weeks of gestation.
2. Subjects with acute bronchiolitis requiring in-patient hospitalization expected to last 24 hours or more.
3. Modified Tal Score (mTal) between 7 to 10 at screening. Note that the oxygen requirement section of the clinical score reflects patient's oxygen saturation without oxygen supplementation.
4. Screening SpO2 of 92% or less in room-air
5. A parent/guardian who is willing to comply with the study procedures and signs an informed consent on behalf of the subject.

Exclusion Criteria:

1. Subjects diagnosed with alveolar pneumonia by chest X-ray and white blood cell (WBC)≥ 15,000/ul and Temp >39°C
2. Previous diagnosis of asthma or cough lasting more than 4 weeks or chronic requirement for asthma medications.
3. Subjects with 2 or more previous physician diagnosed wheezing episodes.
4. Any previous intensive care unit admission for respiratory distress or respiratory-related illness
5. Diagnosis of Bronchopulmonary Dysplasia (BPD) based on medical history and home oxygen use.
6. Subjects on home oxygen use for any reason
7. Presence or use of a nasogastric or orogastric feeding tube
8. Subjects with history of methemoglobinemia, known hereditary methemoglobinemia, and/or methemoglobin >2% for any cause.
9. Use of an investigational drug or device within 30 days before enrollment and/or expected to participate in a new study within 90 days of enrollment.
10. History of frequent epistaxis (>1 episode/month) or significant hemoptysis within 30 days prior to enrollment (≥5 mL of blood in one coughing episode)
11. Taken medications such as chronic systemic corticosteroids, central nervous system (CNS) stimulants, theophylline or aminophylline, anti-arrhythmic within 30 days of screening.
12. Diagnosed with an underlying condition, which significantly affects respiratory system:

    1. Cystic fibrosis (CF), primary ciliary dyskinesia, non-CF bronchiectasis
    2. Immune deficiency
    3. Genetic or neurological disorder capable of causing:

       * Impaired respiratory secretions clearance including insufficient cough
       * chronic respiratory failure and insufficiency
       * restrictive lung disease
    4. Conditions that decrease the muscle strength
    5. Glucose 6-phosphate dehydrogenase deficiency
    6. 6-Phosphogluconate dehydrogenase deficiency
    7. Trisomy 21 (Down Syndrome)
13. Presence of upper airway anomalies that may interfere with breathing, including:

    1. Choanal atresia or stenosis
    2. Cleft lip and palate
    3. Tracheo-esophageal fistula
    4. Tracheal stenosis
    5. Tracheomalacia and/or bronchomalacia
14. History of severe aspiration pneumonia
15. Having the following signs or symptoms:

    1. clinically significant pulmonary (lung) and/or cardiac (heart) congenital malformations
    2. an underlying renal, or liver insufficiency, immunodeficiency, encephalopathy;
    3. known or suspected foreign body aspiration during enrollment.
16. If the first treatment cannot start within 6 hours after signing of the informed consent form (ICF), the subject is not eligible for enrollment.
17. Symptoms (i.e., cough and wheezing) started longer than 72 h before admission to the hospital
18. Per Investigator's discretion, the subject parents/legal guardian(s) are unable to comply with the study procedures.
19. Any reason that, in the opinion of the investigator, may make the subject unfit for this clinical trial.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Time to "fit for discharge" | up to 14 days
  Time to "fit for discharge". "Fit for discharge" is a composite endpoint measured by the following:
  * Achieving Modified Tal score [mTal] ≤ 5 And
  * Oxygen saturation (SpO2) ≥92% at room air (without oxygen supplementation) sustained for at least 2 hours Both of these will be determined from the time of enrollment (when the ICF is signed).

SECONDARY OUTCOMES:
Time to achieve O2 saturation of ≥ 92 %. sustained for at least 2 hours | up to 14 days
  The time in hours calculated from the time of patient's enrollment until the time required to achieve the endpoint.
Hospital Length of Stay (LOS) | up to 14 days
  LOS is measured in hours from the time of patient's enrollment in the study until the physician's order to discharge from the hospital. A patient will be evaluated for discharge from the hospital only after meeting the primary efficacy endpoint.
Modified Tal score [mTal] ≤5 | up to 14 days
  The time in hours calculated from the time of patient's enrollment until the time required to achieve a clinical score of less than or equal to 5.
Incidence of Treatment-Emergent Adverse Events | Baseline to 30 days post dose
  Number of treatment-emergent adverse events (AEs) and Serious AEs

OTHER OUTCOMES:
Admissions to ICU | from enrollment till end of follow up period (30+5 days from enrollment)
  Number of admissions to ICU
Duration of O2 supplementation (in hours) | up to 14 days
  Duration of O2 supplementation (in hours)
Level of O2 supplementation (in %) | up to 14 days
  Level of O2 supplementation (in %)
Nasopharyngeal swab testing for detecting respiratory viruses at baseline and end of treatment | up to 14 days
  Nasopharyngeal swab testing for detecting respiratory viruses at baseline and end of treatment. Will be performed for exploratory purposes only.
Readmission related to bronchiolitis | 30 days from enrollment
  Readmission related to bronchiolitis - percentage of readmissions, related to bronchiolitis within 30 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Goldbart, Principal Investigator — Soroka University Medical Center
Locations (7):
- Israel (7):
  - Haemek Medical Center, Afula
  - Assuta Ashdod, Ashdod
  - Soroka Medical Center, Beersheba
  - Carmel MEdical Center, Haifa
  - Shaarei Zedek Medical Center, Jerusalem
  - Schneider Children's hospital, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldbart A, Lavie M, Lubetzky R, Pillar G, Landau D, Schlesinger Y, Spiegel R, Golan-Tripto I, Nahum A, Greenberg D, Tal A. Inhaled Nitric Oxide for the Treatment of Acute Bronchiolitis: A Multicenter Randomized Controlled Clinical Trial to Evaluate Dose Response. Ann Am Thorac Soc. 2023 Feb;20(2):236-244. doi: 10.1513/AnnalsATS.202103-348OC. PMID 36169967